CLINICAL TRIAL: NCT02886104
Title: Comparison of Hepatectomy and Local Ablation for Resectable Synchronous and Metachronous Colorectal Liver Metastasis (HELARC) ------ a Randomized Controlled Multicenter Clinical Study
Brief Title: Comparison of Hepatectomy and Local Ablation for Resectable Synchronous and Metachronous Colorectal Liver Metastasis
Acronym: HELARC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Second Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2016026
Record Dates: First submitted 2016-08-24; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Secondary Malignant Neoplasm of Liver
Keywords: synchronous; metachronous; colorectal liver metastasis; resection; ablation
MeSH Terms: interventions — Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRLM resection group (Active Comparator): Resection of both primary and secondary tumors in SCRLM and resection of MCRLM. Interventions: Simultaneous resection of both primary and secondary tumors in SCRLM and resection of MCRLM.
  Interventions: Procedure: CRLM resection group
- CRLM ablation group (Experimental): Ablation of CRLM after resection of primary tumor in SCRLM and ablation of MCRLM.
  Interventions: Ablation of liver metastasis within 30 days after resection of primary tumor in SCRLM and ablation of MCRLM.
  Interventions: Device: CRLM ablation group

INTERVENTIONS:
Procedure: CRLM resection group — Simultaneous resection of both primary and secondary tumors in synchronous CRLM or resection of metachronous CRLM.
  Other Names: Hepatectomy
  Arms: CRLM resection group
Device: CRLM ablation group — Microwave ablation of CRLM with a 2.15-gigahertz(GHz) microwave generator and a 14 gauge diameter transcutaneous antenna within 30 days after resection of primary tumor in synchronous CRLM or ablation of metachronous CRLM.
  Other Names: Microwave ablation
  Arms: CRLM ablation group

SUMMARY:
The surgical and local ablation strategy for the treatment of resectable synchronous and metachronous colorectal liver metastases(CRLM) has not still been defined. The purpose of this study is to compare two treatment strategies in which simultaneous resection of both primary and secondary tumor of synchronous CRLM(SCRLM) and resection of metachronous CRLM(MCRLM) is compared with resection of primary tumor and ablation of secondary tumor in SCRLM and ablation of MCRLM. Endpoints include the rate of severe complications and survival.

DETAILED DESCRIPTION:
Colorectal cancer(CRC) kills more than 700,000 patients every year, which is nowadays the world's 3rd common and the 4th deadly tumor. About 50% CRC patients will finally develop colorectal liver metastasis (CRLM). Among the CRLM patients, 20-25% of CRC are found with synchronous colorectal liver metastases (SCRLM) at the first visit. Meanwhile, about 20-30% CRC patients suffer by metachronous colorectal liver metastasis (MCRLM) even after radical resection of primary tumor. It is nowadays admitted that the R0 resection of both primary and secondary tumors in SCRLM and R0 resection of MCRLM represents a feasible and potential curative treatment in patients with resectable CRLM(RCRLM). However, the treatment strategy for some RCRLM (tumor number≤3 and tumor size≤3.0cm), such as whether to choose hepatectomy or local ablation, still remains in debate. In primary hepatocellular carcinoma(HCC), local ablation has been proved to has similar curative effect to that of hepatectomy. Compared to hepatectomy, local ablation has less trauma and more rapid recovery and possible lower hospitalization cost. The curative effect of local ablation is mainly influenced by tumor site and tumor size. On the other side, some RCRLM might develop repeat recurrences even after "R0" resection due to the imaging undetectable micro metastasis. Thus, local ablation might be more suitable for some repeat recurrent CRLM. The aim of this study is to compare the efficacy/safety of local ablation with hepatectomy for RCRLM (tumor number≤3, tumor size≤3.0cm), including both SCRLM and MCRLM. Patients are randomized to CRLM resection group and local ablation group. The primary endpoint is overall survival. Secondary endpoints evaluate the rate of patients with at least one severe complication within 30 days after surgery/ablation and long-term clinical outcomes, in particular disease-free survival.

ELIGIBILITY:
Inclusion Criteria:

1. At least one metastatic adenocarcinoma of liver, histologically proven.
2. At least one adenocarcinoma of colon and/or rectum, histologically proven.
3. No local complication at the time of surgery (no occlusion, no sub-occlusion, no massive hemorrhage, no abscesses or local invasion).
4. No extra-hepatic metastasis.
5. Extra-hepatic disease (EHD) suitable for hepatectomy, liver ablation and anesthesia as long as all sites of EHD disease are radically treated.
6. All the primary and secondary tumors which R0 resections are technically possible. (SCRLM: synchronous resection for both primary and secondary tumors, MCRLM: no local recurrence within 6 months after resection of primary tumor)
7. Residual hepatic volume>30%-40%.
8. At least 2-3 hepatic segments remained after hepatectomy (except S1), residual liver with normal portal vein, hepatic artery and biliary duct, at least 1 of hepatic veins (left, middle and right) not invaded.
9. Tumor size ≤3 cm.
10. Tumor number≤ 3.
11. Tumors located ≥1.0 cm of vulnerable structures, e.g. colon, main trunk of portal vein, hepatic artery, hepatic vein and intrahepatic biliary duct.
12. suitable for both hepatectomy and local ablation after multiple disciplinary team(MDT) discussion.
13. Informed written consent.

Exclusion Criteria:

1. Other malignant tumors history.
2. Complications need emergency surgery (occlusion, sub-occlusion, massive hemorrhage and abscesses, et al.).
3. Colorectal or hepatic tumor extension towards abdominal wall and/or adjacent organ making liver R0 resection impossible immediately.
4. Hepatic lesions diagnosed with ultrasound and MRI making complete ablation impossible immediately.
5. ≤ 2 hepatic segments remained after hepatectomy or residual hepatic volume﹤30%-40%
6. Non resectable lymph node metastasis.
7. American Society of Anesthesiologists(ASA) grading≥ IV and/or Eastern cooperative oncology group(ECOG) score≥ 2. (see appendix)
8. EHD is not recommended.
9. Physical or psychological dependence.
10. Pregnant or breast feeding women.
11. Not controlled preoperational infection.
12. Enrolled in other clinical trials within 4 weeks. Other clinical or laboratorial condition not recommended by investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 548 (Estimated)
Dates: Start 2016-08; Primary Completion 2021-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years

SECONDARY OUTCOMES:
R0 resection rate in both primary and secondary tumor in CRLM | Day of surgery
Death rate during hospitalization or within 30 days after surgery/ablation | 30 days after surgery/ablation
Rate of patients with at least one postoperative severe complication within 30 days after surgery/ablation | 30 days after surgery/ablation
Disease-free survival and 1, 2 and 3-years disease-free survival rate | 1, 2 and 3-years
Complete ablation rate in CRLM | Day of ablation

CONTACTS AND LOCATIONS:
Overall Officials: Meijin Huang, MD,PHD, Principal Investigator — The 6th Affiliated Hospital of Sun Yat-sen University
Locations (1):
- The 6th Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brody H. Colorectal cancer. Nature. 2015 May 14;521(7551):S1. doi: 10.1038/521S1a. No abstract available. PMID 25970450
- [Background] Joranger P, Nesbakken A, Hoff G, Sorbye H, Oshaug A, Aas E. Modeling and validating the cost and clinical pathway of colorectal cancer. Med Decis Making. 2015 Feb;35(2):255-65. doi: 10.1177/0272989X14544749. Epub 2014 Jul 29. PMID 25073464
- [Background] Kopetz S, Chang GJ, Overman MJ, Eng C, Sargent DJ, Larson DW, Grothey A, Vauthey JN, Nagorney DM, McWilliams RR. Improved survival in metastatic colorectal cancer is associated with adoption of hepatic resection and improved chemotherapy. J Clin Oncol. 2009 Aug 1;27(22):3677-83. doi: 10.1200/JCO.2008.20.5278. Epub 2009 May 26. PMID 19470929
- [Background] Bethke A, Kuhne K, Platzek I, Stroszczynski C. Neoadjuvant treatment of colorectal liver metastases is associated with altered contrast enhancement on computed tomography. Cancer Imaging. 2011 Jun 29;11(1):91-9. doi: 10.1102/1470-7330.2011.0015. PMID 21771709
- [Background] Livraghi T. Single HCC smaller than 2 cm: surgery or ablation: interventional oncologist's perspective. J Hepatobiliary Pancreat Sci. 2010 Jul;17(4):425-9. doi: 10.1007/s00534-009-0244-x. Epub 2009 Nov 5. PMID 19890600